CLINICAL TRIAL: NCT00544609
Title: Phase I Trial of Sorafenib in Combination With Radiotherapy in the Treatment of Invasive Bladder Cancer With Conservative Intent
Brief Title: Sorafenib and Radiotherapy in the Treatment of Invasive Bladder Cancer With Conservative Intent
Acronym: SOGUG-07-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-07-01
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Bladder Cancer
Keywords: Bladder; Sorafenib; Radiotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sorafenib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Other): 2 weeks:Sorafenib, 6 weeks and a half:Sorafenib with radiotherapy, 4 weeks:Sorafenib
  Interventions: Drug: Sorafenib; Procedure: Radiotherapy

INTERVENTIONS:
Drug: Sorafenib — Level 1: 200 mg/day Level 2: 400mg/day Level 3: 800mg/day
  Other Names: Nexavar
Procedure: Radiotherapy — 3th-8th week: sorafenib daily with radiotherapy day 1, 2, 3, 4 and 5, 9th week: sorafenib daily with radiotherapy day 1 and 2
  Other Names: Sorafenib; Nexavar

SUMMARY:
Safety profile and to determine maximum tolerated dose of Sorafenib in combination with Radiotherapy in the Treatment of Invasive Bladder Cancer With Conservative Intent

DETAILED DESCRIPTION:
Study phase I in patients with Invasive Bladder Cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with urothelial carcinoma of the bladder, in clinical stages T2-4a N0 M0 (if multifocal evaluation of all lesions by biopsies), who are not candidates for radical cystectomy by medical reasons or refusal.
* No prior treatment with radiotherapy to the bladder or systemic chemotherapy.
* Patients must be ≥ 18 years old.
* Patients must have ECOG performance status 0 to 2.
* Life expectancy of at least 12 weeks.
* Patients with adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

hemoglobin ≥ 9.0 g/dl absolute neutrophil count ≥ 1.500/mm3 platelets ≥ 100.000/mm3. total bilirubin ≤ 1.5 times the upper limit of normality SGOT (AST) and/or SGPT (ALT) ≤ 2.5 times the upper limit of normality alkaline phosphatase ≤ 4 x ULN serum creatinine ≤1.5 upper limit of normality PT-INR/PTT < 1.5 x upper limit of normality creatinine clearance ≥ 40 ml/min using Cockcroft-Gaul

* Patients must give their written informed consent before any procedure related to the study is performed; therefore, it must be given at the selection visit. The patient must be informed that he has the right to withdraw from the study at any time, without any kind of prejudice.
* Patients who are capable of accomplishing the study's requirements and without any impediments to follow the instructions.
* Women of fertile age must have a negative result in the pregnancy test performed 7 days before the beginning of the administration of the study medication.
* Patients from both sexes must use adequate contraceptive methods (oral or injectable contraceptives, intrauterine device, condom, sterilization) whilst participating in the protocol. After the retreat of treatment with sorafenib, the contraceptive methods must be used during 4 weeks in women and during 3 months in men.

Exclusion Criteria:

* Patients with active infection or other serious medical conditions (autologous bone marrow transplant or stem cell rescue within 4 months of study, patients undergoing renal dialysis, known HIV infection or chronic hepatitis B or C, active clinically serious infections > CTCAE Grade 2, non-healing wound, ulcer, or bone fracture).
* Abuse of substances, clinical conditions, psychological or social, that would preclude appropriate informed consent or compliance with protocol.
* Concurrent treatment with other experimental drugs (within 30 days prior to study entry).
* Concurrent treatment with other anti-cancer- or immunotherapy during the study or within 4 weeks of study entry.
* Treatment wuth mitomycin C or nitrosureas during 6 weeks prior of study entry.
* History of prior malignancies within the preceding 5 years other than previously treated basal cell carcinoma of the skin, incipient prostate cancer and in situ cervix carcinoma.
* Pregnant or breast feeding patients.
* Known or suspected allergy to sorafenib.
* Cardiac disease: Congestive heart failure > class II NYHA; active CAD (myocardial infarction more than 6 months to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy (beta blockers or digoxin are permitted).
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management.
* Known brain metastasis. Patients with neurological symptoms should undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Patients with hydronephrosis.
* Patients with seizure disorder requiring medication (such as steroids or antiepileptics).
* History of organ allograft.
* Patient unable to swallow oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety profile of Sorafenib in combination with Radiotherapy. | 12 weeks
Maximum tolerated dose of Sorafenib in combination with Radiotherapy. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xavier García del Muro Solans, MD, Study Chair — Institut Català d' Oncología, Barcelona; Salvador Villà Freixa, MD, Study Chair — Institut Català d' Oncología, Barcelona
Locations (3):
- Spain (3):
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Català d' Oncología, Barcelona